CLINICAL TRIAL: NCT07245719
Title: Stryker Universal Midface and Upper-Face Fixation System: A Retrospective Post Market Follow Up to Confirm Safety, Performance and Effectiveness of The Universal CMF System
Brief Title: Stryker Universal Midface and Upper-Face Fixation System: A Retrospective Post Market Follow Up
Acronym: UMF
Status: Recruiting | Type: Observational
Sponsor: Stryker Craniomaxillofacial (Industry)
Responsible Party: Sponsor
Other Study IDs: Universal CMF System _2023_01
Record Dates: First submitted 2025-08-07; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Zygomatic Fractures; Orbital Fractures; Maxilla Fractures; Facial Fractures
MeSH Terms: conditions — Zygomatic Fractures; Orbital Fractures; Maxillary Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Upper-Face and/or Mid-Face modules (1.2 / 1.7 modules) of the Stryker Universal CMF System — The Universal CMF System is a plate and screw system intended for osteotomy, stabilization, and rigid fixation of CMF fractures and reconstruction.
  Depending on the selected module, the design of the devices is more suitable for specific indications within the broad indication of CMF fractures and CMF reconstructive surgeries.

SUMMARY:
A retrospective post-market clinical follow-up to confirm the performance and safety of the Upper-Face and Mid-Face modules of the Stryker Universal CMF System in a clinical setting. The study is performed to confirm the product's performance and safety by systematically collecting clinical data on its use.

DETAILED DESCRIPTION:
This is a retrospective non-interventional post-market follow up aiming at confirming safety and performance of the Stryker Universal System when used in a clinical setting. This study will include patients who have previously undergone a surgical procedure involving the Study Device, with surgical outcomes evaluated retrospectively. Based on a non-inferiority study power calculation a minimum of 120 patients will be enrolled in the study. Additional patients may be enrolled up to 150 subjects depending on site enrolment rate and patient availability. Up to 2 investigational sites within the United States will participate in this study. The primary outcome parameter evaluating successful stabilization and/or fixation of bony segments without the need for unplanned revision surgery will be evaluated at all available follow-up timepoints of the included patients.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature patients at the time of surgery.
2. Patients who underwent a craniomaxillofacial procedure using implants of the Upper-Face and/or Mid-Face modules (1.2 / 1.7 modules) of the Stryker Universal CMF System as per routine clinical practice.
3. Patients for whom data on the primary outcome variable is available.
4. Patients with data available from follow-up visits.

Exclusion Criteria:

1. Patients with active infections at the time of surgery.
2. Patients with known metal allergies and/or foreign body sensitivity at the time of surgery.
3. Subjects with non-reducible and unstable fractures (except reconstruction plates) at the time of surgery that were treated with the subject devices.
4. Patients who underwent secondary reconstructions with non-secondary reconstruction plates
5. Patients with limited blood supply or insufficient quality or quantity of bone at the time of surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified as having had a surgical procedure involving the Subject Device.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Successful stabilization and/or fixation of bony segments without the need for unplanned revision surgery | Data collected at a single time point per patient in the course of 12 months.
  Assessed by reviewing adverse events in patient medical charts at time point after surgery. Used to document whether an unplanned revision surgery was required or not for patients.

SECONDARY OUTCOMES:
Intraoperative complications | Data collected at a single time point per patient in the course of 12 months.
  Determined by intraoperative adverse events reported from patient medical charts.
Postoperative complications | Data collected at time points per patient in the course of 12 months.
  Determined by post operative adverse events reported from patient medical charts.
Any known adverse events potentially related to the primary outcome objective and/or device | Data collected at time points per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Implant failure | Data collected at time points point per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Operating room (OR) time | Data collected at a single time point per patient in the course of 12 months.
  Time patients are operated (dd:hh)
Hospitalization time | Data collected at a single time point per patient in the course of 12 months.
  Time the patient was hospitalized post procedure (ICU and normal ward; dd:hh)
Post-operative bone consolidation | Data collected at time points point per patient in the course of 12 months.
  Clinical observation of post-op bone consolidation (medical charts) Timing of post-op observation of bone consolidation (yymmdd) Availability of post op imaging to determine bone consolidation Timing of post-op imaging (number of scans, yymmdd)

OTHER OUTCOMES:
Age | Data collected at a single time point per patient in the course of 12 months.
  Patient age (year of birth, age in years)
Primary indication for the surgery / diagnosis | Data collected at a single time point per patient in the course of 12 months.
  Diagnosis collected from patient medical charts
Surgical approach/access | Data collected at a single time point per patient in the course of 12 months.
  Surgical approach taken for the procedure. Including: orthognathic, trauma, oncological, congenital defect, other. Usage of the device in the maxilla and maximal incisal mouth opening (post- and pre-operation). Application of post-operative Maxillo-Mandibular Fixation
Anatomical area treated | Data collected at a single time point per patient in the course of 12 months.
  Area to treated by the device: orbital region, zygomatic region, dento-alveolar region, maxilla, frontal region, other.
Other implants used | Data collected at time points per patient in the course of 12 months.
  Other implants that may have been used during the surgical procedure.
Max follow-up time | Data collected at a single time point per patient in the course of 12 months.
  Maximum post operative follow up time for patients within standard of care. Reported in patient medical charts during hospital follow up visits.
Orthognathic cases | Data collected at a single time point per patient in the course of 12 months.
  Satisfactory occlusion expected to be achieved after potential additional orthodontic treatment.
Patient Radiation Exposure | Data collected at time points per patient in the course of 12 months.
  Exposure of patient to radiation therapy within 12 months around the surgery date recorded in patient medical charts (number and type of radiation procedures performed). Radiation therapy performed on the anatomical area treated with the device. Any postoperative radiation therapy recorded in patient medical charts.
Sterilization method used | Data collected at a single time point per patient in the course of 12 months.
  Sterilization method used for the device. Qualitative responses from site.
Tightening of screws | Data collected at a single time point per patient in the course of 12 months.
  Tools used to fix the device during the procedure. Manually, electric screw driver
Implants Used | Data collected at a single time point per patient in the course of 12 months.
  Quantity, part numbers & descriptions of implants used from the device.
Gender | Data collected at a single time point per patient in the course of 12 months.
  Patient gender (Male, Female, undifferentiated, unknown)
Height | Data collected at a single time point per patient in the course of 12 months.
  Patient height (cm, feet, inches)
Weight | Data collected at a single time point per patient in the course of 12 months.
  Patient weight (kg, lb)
Year smoking was stopped | Data collected at time points per patient in the course of 16 months.
  Year smoking was stopped (YYYY)
Smoking frequency | Data collected at time points per patient in the course of 12 months
  The frequency of exposure to smoking during periods of smoking (average number of cigarettes per day).
Smoking duration | Data collected at time points per patient in the course of 12 month
  Duration of smoking (pack years)
Years of active smoking | Data collected at time points per patient in the course of 12 months
  Total number of years active smoker (YY)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medicine Oral and Maxillofacial Surgery 525 East 68th Street, F-2132, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided